CLINICAL TRIAL: NCT06390735
Title: Effectiveness of a Web-based Psychoeducation on Antenatal Depression Help-seeking in Eswatini
Brief Title: Antenatal Depression Help-seeking Trial in Eswatini
Acronym: ADHS-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Lindelwa Portia Dlamini, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N202312058; EHHRRB 194/2023 (Other: Eswatini Health and Human Research Review Board)
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Help-Seeking Behavior; Help-seeking Intention; Antenatal Depression
Keywords: antenatal depression; Web-based interventions; Psychoeducation; RCT; Eswatini; Help-seeking
MeSH Terms: conditions — Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: This two armed trial will include an intervention group and a waitlist control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mommy ReachOut intervention (Experimental): The intervention group will receive the Mommy ReachOut intervention, which is a web-based psychoeducation, consisting of a total of 4 sessions to be released over a 2-week period. Two sessions will be released each week, with each session consisting of readable mental health information and videos. Content for this intervention was based on previous reviews, previous intervention studies and the Diagnostic and Statistical manual of mental health disorders (DSM-5). Session content included basic information about antenatal depression, shared antenatal depression experiences, issues around stigma towards antenatal depression, and local resources available for antenatal women with depression in Eswatini.
  Interventions: Behavioral: Mommy ReachOut Intervention
- waitlist control (No Intervention): Participants in the control group will have access to the active treatment after completing the 6-week waiting period. Once the control participants complete the 1-month follow-up assessment, they will receive a website link to access the complete Mommy ReachOut intervention.

INTERVENTIONS:
Behavioral: Mommy ReachOut Intervention — The momy reachOut intervention is a web-based psycho-education with 4 sessions, released over a two week period.
  Arms: Mommy ReachOut intervention

SUMMARY:
The goal of this trial to test if a web-based psychoeducation will work in improving depression help-seeking intention and behavior among antenatal women with probable depression in Eswatini. The main question it aims to answer is:

• Does the web-based psychoeducation improve depression help-seeking intention and help-seeking behavior in antenatal women with probable depressive symptoms?

Researchers will compare this web-based psychoeducation to a waitlist control, to see if the program works in improving depression help-seeking intention and behavior during pregnancy.

* The psychoeducation program will have a total of 4 sessions, which will be given to participants over a two-week period. two sessions will be delivered each week.
* Participants will be asked questions before the intervention starts, immediately the intervention ends as well as after a month of completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Less than 30 weeks of gestation,
* Aged 18 or above
* With probable depression (Edinburg Postnatal depression scale; EPDS > 10)
* Has access to a smart phone
* Fluent in spoken and written Siswati or English (with at least secondary school education)
* Planning to remain in the country for the next 2 months
* Willing to share her dominant phone number with the study team
* Willing to participate in the intervention study

Exclusion Criteria:

* Antidepressants or other depression treatments
* Currently enrolled in another trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Help-seeking Intention | Baseline; Immediately post intervention; follow-up at 1 month post intervention
  General Help Seeking Questionnaire - This 9 item scale adopted a 3 point Likert scale (Unlikely, maybe, Likely) to measure help-seeking intention. The total score is computed by summing up all item scores, where a higher score indicates higher help-seeking intention. The total possible score ranges from 9 to 27.
Help-seeking Behavior | Baseline; Immediately post intervention; follow-up at 1 month post intervention
  Actual Help Seeking Questionnaire - This 9 item scale uses binary responses (Yes or No) to measure actual help-seeking behavior. The total score is computed by summing up all item scores, where a higher score indicates higher help-seeking behavior. The total possible score ranges from 0 to 9.

SECONDARY OUTCOMES:
Antenatal depressive symptoms | Baseline; Immediately post intervention; follow-up at 1 month post intervention
  Edinburgh Postnatal Depression Scale - A set of 10 items are used to measure antenatal depressive symptoms on a 4-point Likert scale (0-3). The overall score ranges from 0 to 30 and is computed by summing up all item scores. A high sum of scores indicates a high level of depressive symptoms.
Health belief | Baseline; Immediately post intervention; follow-up at 1 month post intervention
  Theory of Planned Behavior questionnaire - The tool has 13 items that rate the constructs of the theory of planned behavior on a 5-point Likert scales (strongly disagree to strongly agree). The possible score ranges from 13 to 65, with higher scores indicating more favorable attitudes towards help-seeking, greater subjective norms to seek help, and more control over one's behavior.
Antenatal depression Stigma | Baseline; Immediately post intervention; follow-up at 1 month post intervention
  Depression stigma scale - The 9 items in this scale measure personal stigma towards depression. Responses to each item are measured on a five-point Likert scale (strongly disagree to strongly agree). The total score is through summing up all item scores and a total possible score ranges from 0 to 36. A higher score indicates higher levels of personal depression stigma
Depression literacy | Baseline; Immediately post intervention; follow-up at 1 month post intervention
  Depression literacy scale - The scale measures participants knowledge of the signs of depression, risk factors, and treatment among others. participants respond to each item with a true (1) or false (0), therefore, the total possible score ranges from 0 to 22. From summing up all item scores, a higher score will indicate high antenatal depression literacy.

CONTACTS AND LOCATIONS:
Locations (2):
- Eswatini (2):
  - Mbabane Government Public Health Unit, Mbabane, Hhohho Region
  - King Sobhuza II Public Health Unit, Manzini

IPD SHARING:
Plan to Share IPD: No